CLINICAL TRIAL: NCT03864627
Title: A Randomized, Double-blind, Placebo-controlled, Multicentre Phase 2 Study to Evaluate the Safety and Tolerability of Subcutaneous MOR106 Administered Concomitantly With Topical Corticosteroids for Eight Weeks, in Adult Subjects With Moderate to Severe Atopic Dermatitis
Brief Title: A Study to Evaluate the Safety and Tolerability of MOR106 Administered Concomitantly With Topical Corticosteroids, in Adult Participants With Moderate to Severe Atopic Dermatitis
Acronym: GECKO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: MOR106 clinical development in atopic dermatitis was stopped for futility
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MOR106-CL-204
Record Dates: First submitted 2019-03-05; First posted 2019-03-06 (Actual); Results first posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants will receive MOR106 matching placebo via s.c. injection every other week on Day 1, 15, 29 and 43 given concomitantly with a medium potency TCS once daily until Day 57.
  Interventions: Drug: Placebo
- MOR106 320 mg (Experimental): Participants will receive MOR106 320 milligrams (mg) via s.c. injection every other week on Day 15, 29 and 43 given concomitantly with a medium potency topical TCS once daily until Day 57. A loading dose of MOR106 2 x 320 mg via s.c. injection will be administered on Day 1.
  Interventions: Drug: MOR106

INTERVENTIONS:
Drug: MOR106 — MOR106 liquid formulation for s.c. injection administered concomitantly with TCS (medium potency).
  Arms: MOR106 320 mg
Drug: Placebo — Placebo liquid formulation for s.c. injection administered concomitantly with TCS (medium potency).
  Arms: Placebo

SUMMARY:
To investigate the safety and tolerability of repeated subcutaneous (s.c.) doses of MOR106 administered concomitantly with topical corticosteroids (TCS) in participants with moderate to severe atopic dermatitis (AD) who are candidates for systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

* A BMI 18 - 40 kilogram per meter square (kg/m^2), inclusive.
* Diagnosis of atopic dermatitis for at least one year since first diagnosis as per the Hanifin and Rajka Criteria.
* Eczema Area and Severity Index (EASI) ≥ 16 at the screening and at the baseline visit (Day 1 predose).
* Investigators' Global Assessment (IGA) score ≥ 3 (on the 0 to 4 IGA scale, in which 3 is moderate and 4 is severe) at the screening and baseline visits.
* Greater than or equal to 10% body surface area (BSA) of AD involvement at the screening and baseline visits.
* Willingness to use a non-medicated, simple bland emollient twice daily for at least 7 days before the baseline visit and throughout the study.

Exclusion Criteria:

* Prior treatment with MOR106.
* Known hypersensitivity to any investigational medicinal product (IMP) ingredients as determined by the investigator (such as, but not limited to, anaphylaxis requiring hospitalization).
* AD lesions located predominantly (≥ 50% of cumulative lesional area) on face and genital areas.
* Any concurrent illness, condition, disability, or clinically significant abnormality (including laboratory tests, a New York Heart Association Classification (NYHA) ≥ III/IV) or clinically significant illness in the 3 months prior to initial IMP administration that, in the investigator's opinion, represents a safety risk for the participant's participation in the study, may affect the interpretation of clinical safety or efficacy data, or may prevent the participant from safely completing the assessments required by the protocol.
* Clinically significant abnormalities at the discretion of the investigator detected on vital signs or physical examination (other than AD) at screening or baseline (Day 1 predose).
* History of or a current immunosuppressive condition (e.g. human immunodeficiency virus [HIV] infection, as determined by a positive HIV test at screening).
* Active chronic or acute skin infection requiring treatment with systemic (oral, sc or iv) antibiotics, antivirals or antifungals within 4 weeks of baseline, or clinical signs of infective eczema within 7 days before baseline (Day 1 pre-dose).
* Having used any of the following treatments:

  * Prior exposure to Dupilumab.
  * Immunosuppressive/immunomodulating drugs (e.g. systemic corticosteroids, cyclosporine, mycophenolate-mofetil, interferon (IFN)-γ, azathioprine, methotrexate) within 4 weeks of baseline (Day 1) visit.
  * Phototherapy (ultraviolet B [UVB] or Psoralen Ultraviolet A [PUVA]) for AD within four weeks of baseline (Day 1) visit.
  * Treatment with TCS or topical calcineurin inhibitor (TCI) within 7 days before the baseline (Day 1) visit.
  * Treatment with biologics within five half-lives (if known) or 12 weeks prior to baseline visit, whichever is longer.
  * Regular use (more than two visits per week) of a tanning booth/parlor within 4 weeks of the baseline visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Galapagos Medical Information, Study Director — Galapagos NV
Locations (14):
- United States (14):
  - First OC Dermatology, Fountain Valley, California
  - Marvel Research, LLC, Huntington Beach, California
  - LA Universal Research Center, Inc., Los Angeles, California
  - MedDerm Associates, San Diego, California
  - Encore Medical Research, Hollywood, Florida
  - Advanced Research Institute of Miami LLC, Homestead, Florida
  - Vista Health Research, Miami, Florida
  - Arlington Dermatology, Rolling Meadows, Illinois
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - DS Research, Louisville, Kentucky
  - Greenwich Village Dermatology, New York, New York
  - Center for Clinical Studies, Houston, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Center for Clinical Studies, Webster, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States. The first participant was screened on 25 Mar 2019. The last study visit occurred on 27 Feb 2020.
Pre-assignment Details: A total of 76 participants were screened of which 33 participants were randomized into the study.
Groups:
- Placebo: Participants received MOR106 matching placebo via subcutaneous (s.c.) injection every other week on Day 1, 15, 29 and 43 given concomitantly with medium potency topical corticosteroid (TCS) once daily until Day 57.
- MOR106 320 mg: Participants received MOR106 320 milligrams (mg) via s.c. injection every other week on Day 15, 29 and 43 given concomitantly with a medium potency TCS once daily until Day 57. A loading dose of MOR106 2 x 320 mg via s.c. injection was administered on Day 1.
Period: Overall Study
Arm/Group | Placebo | MOR106 320 mg
Started | 11 | 22
Completed | 7 | 10
Not Completed | 4 | 12
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 4 | 8
Not completed — Study terminated by sponsor | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who received at least one dose of investigational medicinal product (IMP).
Groups:
- Placebo: Participants received MOR106 matching placebo via s.c. injection every other week on Day 1, 15, 29 and 43 given concomitantly with medium potency TCS once daily until Day 57.
- MOR106 320 mg: Participants received MOR106 320 mg via s.c. injection every other week on Day 15, 29 and 43 given concomitantly with a medium potency TCS once daily until Day 57. A loading dose of MOR106 2 x 320 mg via s.c. injection was administered on Day 1.
- Total: Total of all reporting groups
Arm/Group | Placebo | MOR106 320 mg | Total
Number analyzed (Participants) | 11 | 22 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.8 (17.85) | 36.1 (13.34) | 37.4 (14.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 18
  Male | 4 | 11 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 11 | 16
  Not Hispanic or Latino | 6 | 11 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 5 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 9 | 15 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Adverse Event of Special Interest (AESIs), Serious Adverse Events (SAEs)
Description: An Adverse Events (AE) was any untoward medical occurrence, new or worsening of any pre-existing condition, in a clinical study participant administered a medicinal product and which did not necessarily had to have a causal relationship with the treatment. TEAEs: AES with an onset date on or after the start date of the IMP administration. AESIs: skin-related events (SRE) (except exacerbation and infective exacerbation of AD) or injection site reactions (ISRs) as per common terminology criteria for AEs (Grade 3: ulceration or necrosis; severe tissue damage; operative intervention indicated, Grade 4: life-threatening consequences; urgent intervention indicated, Grade 5: death ). An SAE: AE that resulted in any of the following outcomes: death; life threatening; results in persistent or significant disability/incapacity; requires in-patient hospitalization or prolongation of existing hospitalization; congenital anomaly/birth defect; is medically significant.
Time Frame: Day 1 up to Day 169/Early discontinuation(ED)
Population: The safety analysis set included all participants who received at least one dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MOR106 320 mg
Number analyzed (Participants) | 11 | 22
Participants
  TEAE | 5 | 11
  AESI: SRE | 2 | 1
  AESI: ISRs | 0 | 0
  SAE | 0 | 1

2. Secondary Outcome: Serum Concentrations of MOR106
Time Frame: Day 1, Day 4, Day 15, Day 29, Day 43, Day 57, Day 71, Day 85, Day 99, Day 113, Day 127, Day 141, Day 155 and Day 169
Population: The pharmacokinetic (PK) analysis population was a subset of safety analysis set and included all participants who had available and evaluable serum concentration data. Participants in PK population with available data at specified timepoint.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (µg/mL)
Arm/Group | MOR106 320 mg
Number analyzed (Participants) | 20
microgram per milliliter (µg/mL)
  Day 1 | 0.149 (0.2505)
  Day 4: number analyzed (Participants) | 18
  Day 4 | 61.150 (28.3850)
  Day 15: number analyzed (Participants) | 18
  Day 15 | 41.278 (21.4046)
  Day 29: number analyzed (Participants) | 15
  Day 29 | 39.473 (15.8087)
  Day 43: number analyzed (Participants) | 10
  Day 43 | 42.537 (23.8095)
  Day 57: number analyzed (Participants) | 11
  Day 57 | 40.934 (17.6737)
  Day 71: number analyzed (Participants) | 9
  Day 71 | 16.593 (7.3308)
  Day 85: number analyzed (Participants) | 6
  Day 85 | 9.775 (3.2489)
  Day 99: number analyzed (Participants) | 6
  Day 99 | 5.092 (1.0801)
  Day 113: number analyzed (Participants) | 6
  Day 113 | 2.415 (1.3466)
  Day 127: number analyzed (Participants) | 9
  Day 127 | 1.407 (0.8124)
  Day 141: number analyzed (Participants) | 7
  Day 141 | 1.812 (2.4765)
  Day 155: number analyzed (Participants) | 6
  Day 155 | 1.043 (1.2149)
  Day 169: number analyzed (Participants) | 7
  Day 169 | 0.690 (0.9707)

3. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADAs)
Time Frame: Day 1 up to Day 169/ED
Population: Safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MOR106 320 mg
Number analyzed (Participants) | 11 | 22
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 169/ED
Description: Safety analysis set.
Arm/Group | Placebo | MOR106 320 mg
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/11 | 1/22
Other Adverse Events (participants affected / at risk) | 5/11 | 11/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=11) | MOR106 320 mg (N=22)
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=11) | MOR106 320 mg (N=22)
Injection site reaction (General disorders) | 1 | 2
Folliculitis (Infections and infestations) | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Burning sensation (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Atrioventricular block first degree (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated as MOR106, clinical development in atopic dermatitis was stopped for futility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must review and approve any results of the study or abstracts for professional meetings prepared by the investigator(s). Published data must not compromise the objectives of the study. Data from individual study centers in multicenter studies must not be published separately.

DOCUMENTS (2):
  • Study Protocol (2019-06-25): https://cdn.clinicaltrials.gov/large-docs/27/NCT03864627/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-12): https://cdn.clinicaltrials.gov/large-docs/27/NCT03864627/SAP_001.pdf